CLINICAL TRIAL: NCT04024397
Title: Unintended Prolonged Opioid Use
Brief Title: A Study to Evaluate Unintended Prolonged Opioid Use
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, W. Michael Hooten, Principal Investigator, Mayo Clinic
Other Study IDs: 18-010484; U01TR002743 (NIH)
Record Dates: First submitted 2019-07-11; First posted 2019-07-18 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Opioid Use

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Researchers are trying to better understand how people who are prescribed opioids for short-term use, go on to receive this type of medication on a longer-term basis.

DETAILED DESCRIPTION:
Identify incident cases of UPOU and prospectively assess their characteristics in comparison to new opioid users who do not progress to UPOU. At each site, opioid-naïve adults who receive opioid prescriptions will be enrolled. Opioid prescriptions (both written and filled) and self-reported opioid use will be followed, and those subjects progressing to UPOU will be identified in real time. Matched samples of patients who do and do not develop UPOU will be recruited for assessment of framework elements related to patient characteristics,including biochemical confirmation of opioid use, pain-related measures (including psychological variables), and medical and social histories. Using the information gathered in Aim 1, structural equation modeling will be utilized to evaluate the associations UPOU and the patient domain.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* No use of opioids for 6 months prior to the issuance of the initial opioid prescription
* Willingness to participate in all aspects of the study including use of the Hugo platform on their personal smartphone

Exclusion Criteria:

* Cancer-associated pain
* Concurrent treatment for cancer (e.g., chemotherapy, radiation therapy)
* Residence in an extended care facility
* Any operation or hospitalization within the past 6 months
* Mental health disorders that could impede functioning in an ambulatory care setting (e.g., schizophrenia, dementia)
* Non-English speaking individuals
* No smartphone
* Use of a pharmacy that is not compatible with the Hugo platform.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any individual that receives an opioid prescription.
Sampling Method: Non-Probability Sample
Enrollment: 1796 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Assess the rate of long-term opioid use | Six months
  At month 6 following the receipt of the initial opioid prescription, the status of opioid use will be assessed to determine the rate of converting to long-term use.

SECONDARY OUTCOMES:
Assess patient factors associated with development of long-term opioid use | Six months
  Patient factors potentially associated development of long-term opioid use will be assessed including depressive symptoms as measured using the Center for Epidemiological Studies-Depression Scale. Scores on the scale range from 0 to 60 where higher scores indicated greater levels of depression. A cut-off score of 27 or greater indicates clinically significant levels of depression.

CONTACTS AND LOCATIONS:
Overall Officials: W. Michael Hooten, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hooten WM, Erickson DJ, Chawarski M, Scholz NA, Waljee JF, Brummett CM, Jeffery MM. Unintended Prolonged Opioid Use: Protocol for a Case-Controlled Trial. JMIR Res Protoc. 2025 Mar 24;14:e72032. doi: 10.2196/72032. PMID 39992690
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials